CLINICAL TRIAL: NCT06441071
Title: Effect of Different Patient's Positions on Postoperative Analgesia of Ultrasound-guided Erector Spinae Plane Block
Brief Title: Patients' Positions on Analgesic Efficacy of ESPB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KY20240419-03
Record Dates: First submitted 2024-05-08; First posted 2024-06-04 (Actual); Last update posted 2025-07-21 (Actual); Status verified 2025-03

CONDITIONS: Erector Spinae Plane Block
Keywords: Paravertebral thoracic block; Clinical application; Perioperative analgesia; Erector spinae plane block
MeSH Terms: interventions — Patient Positioning

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group S (Experimental): After completion of the erector spinae plane block, patients in group S remained in the supine position for 30 minutes.
  Interventions: Procedure: position
- Group L (Experimental): After completion of the erector spinae plane block, patients in group L remained in the lateral position for 30 minutes.
  Interventions: Procedure: position
- Group P (Experimental): After completion of the erector spinae plane block, patients in group P remained in the prone position for 30 minutes.
  Interventions: Procedure: position
- Group C (Other): After completion of the paravertebral block, patients in group C remained in the supine position for 30 minutes.
  Interventions: Procedure: position

INTERVENTIONS:
Procedure: position — Patients undergoing Video-assisted Thoracoscopic Surgery were selected for the study, and nerve block was performed before surgery, followed by holding different positions for 30 min, after which the effect of the block was measured.

SUMMARY:
The goal of this clinical trial is to learn if patients remaining different positions for 30min after receiving ultrasound-guided erector spinae plane block influenced the postoperative analgesia. The main questions it aims to answer are:

Does patients maintain prone position or lateral position for 30 min after ESPB provided superior analgesic effect than in the supine position? Is ESPB not inferior to PVB considering postoperative opioid consumption ? Researchers will compare the opioid consumption 24h postoperatively among the patients remaining supine, lateral, prone position after ESPB and PVB to see if patients maintaining lateral or prone position provided excellent postoperative analgesia.

Participants will:

Maintaining supine lateral or prone position for 30 min following ESPB or receiving PVB.

Receiving postoperative NRS and QoR assessment

DETAILED DESCRIPTION:
After signed the informed consent form, 200 patients scheduled for elective thoracoscopic surgery were randomly divided into four groups: supine position group (group S, n = 50), prone position group (group P, n = 50), lateral position group (group L, n = 50) and paravertebral block group (group C, n = 50). After ESPB block, the corresponding position was maintained for 30 minutes.

Ultrasound-guided ESPB was performed 30min before general anesthesia. Ultrasound-guided ESPB methods: The ultrasonic high-frequency linear array probe (5-13 MHZ, Sonosite, USA) was placed parallel to the spine on the surface of the transverse process tip of the seventh thoracic vertebra. Under ultrasound, the transverse process and the surface of the erector spinae were clearly exposed. Then a long beved-plane needle was used, and the needle was inserted from the head side. 2ml of normal saline was injected using the water separation technique to confirm the position of the needle tip, and then 30ml 0.375% ropivacaine was injected.

After completion of the block, patients in group S were kept in the supine position for 30min, patients in group L were kept in the upper lateral position for 30min, and patients in group P were kept in the prone position for 30min. After 30 minutes of observation, an anesthesiologist who was unaware of the grouping used an ice cube to determine the extent of sensory block. General anesthesia was then performed.

General anesthesia was performed as follows: routine ECG monitoring was performed after the patient was admitted to the operating room, and invasive arterial blood pressure was monitored by radial artery puncture and catheterization. General anesthesia was induced with dexamethasone 10mg, midazolam 0.05mg.kg-1, propofol 1.5-2.0 mg.kg-1, sufentanil 0.2 ug.kg-1, cisatracurium 0.2 mg.kg-1, and then a double-luminal bronchial tube was inserted under a video laryngoscope and mechanically ventilated (tidal volume: 6-10ml.kg-1,PEEP: 3-5 cm H2O). Anesthesia was maintained with propofol (2-4 mg.kg-1.h-1), remifentanil (0.12-0.3 ug.kg-1.min-1) and Micuronium (0.6mg.kg-1.h-1). Intraoperative hemodynamics was maintained within 20% of baseline. Flurbiprofen axetil 50mg was given intravenously for analgesia and tropisetron 4mg was given to prevent nausea and vomiting when there were no contraindications during the operation. Oxycodone 3mg was administered intravenously 30min before the end of the procedure. At the end of the operation, the patient was transferred to PACU with an endotracheal tube. After neuromuscular blocking antagonism, the tracheal tube was extubated.

NRS was used to evaluate the pain scores at rest and during movement at 1, 3, 6, 12 and 24h ，48h after operation by a nurse who was unaware of the grouping. Oxycodone 30mg diluted to 150ml was used for patient-controlled intravenous analgesia after operation. The parameters of analgesia pump were set as background dose 0.5 ml.h-1, bolus 5ml, lockout time 8min. If NRS≥4 at rest after surgery, patient-controlled analgesia (PCA) was performed by pressing the PCA pump. When NRS≥4 at rest was still ≥4 after two times of PCA, oxycodone 1mg was given once as rescue analgesia, and the patients were reevaluated until NRS≤3.

ELIGIBILITY:
Inclusion Criteria:

Patients undergoing Video-assisted Thoracoscopic Surgery under elective general anaesthesia were selected, regardless of sex, age 18-80 years, BMI: 18-30 kg.m-2, ASA classification I-III.

Exclusion Criteria:

1. Allergy to the study drug or allergy to local anaesthetics;
2. History of opioid abuse;
3. Previous nerve block puncture with puncture site infection；
4. Peripheral neuropathy；
5. Coagulation abnormalities, defined as prothrombin time or partial activation time prothrombin time exceeding standard values or international normalised ratio (INR) ≥ 1.4, or platelet count ≤ 70 x 109 L-1.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-06-14 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative Oxycodone dosage | 24 hour postoperatively
  Cumulative oxycodone dosage 24 hour postoperatively

SECONDARY OUTCOMES:
Loss to cold sensation of skin | 30 minute after block
  The sensation to cold was assessed with ice. The area include the anterior chest wall (midclavicular line), lateral chest wall (posterior axillary line), and posterior chest wall (paraspinal zone) by a researcher who was blinded to group allocation.
NRS(Numeric Rating Scales) score | Postoperative 1, 3, 6, 12, 24, 48 hour
  Postoperative 1, 3, 6, 12, 24, 48 hour NRS (Numeric Rating Scales) score. Numerical Rating Scale (NRS): This scale is composed of 11 numbers from 0 to 10, with higher numbers increasing the severity of pain.
Adverse reaction | 24, 48 hour postoperatively
  This includes dizziness, nausea, vomiting, etc.
QoR-15 score(Quality of Recovery,QoR) | Day 1 and 2 postoperatively
  Postoperative QoR-15(Quality of Recovery) score was used to evaluate the quality of early postoperative recovery on postoperative day 1 and 2. . The QoR-15 score(Quality of Recovery,QoR) included 5 dimensions including emotional state, physical comfort, psychological support, physical independence and pain, with a total of 15 items. Each item scored from 0 to 10, with higher scores being better.
Opioid dosage | 1, 3, 6, 12, 24, 48 hour postoperatively
  Postoperative opioid consumption dosage.
Patient Comfort Scale score | 30 minute after block
  used to assess the comfort level of the patient according to the position during the procedure (grade 0=help, 2=uncomfortable, 4=mild discomfort, 6=feeling OK, 8=pretty comfortable, and 10=feeling great)
Hemodynamic profile | Heart rate changes before blockade, 5minute after blockade, 10 minute after blockade, 20minute after blockade, 30minute after blockade
  Hemodynamic changes(Heart rate ) during blockade procedure
Hemodynamic profile | Mean arterial pressure changes before blockade, 5minute after blockade, 10 minute after blockade, 20minute after blockade, 30minute after blockade
  Hemodynamic changes(Mean arterial pressure ) during blockade procedure

CONTACTS AND LOCATIONS:
Overall Officials: Tao Shan, Study Director — Nanjing First Hospital, Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No